CLINICAL TRIAL: NCT03977064
Title: Fertility and Cardiovascular Risk in Men With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EK205/16
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will receive pseudonymous data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive treatment group (Experimental): The intensive treatment group will pass a life-style intervention program including consequent escalation of measures to reach sustained reduction of 10% of initial body weight at minimum.
  Interventions: Behavioral: Life style change and weight reduction
- Standard treatment group (No Intervention): Patients will be taken care of by general physician without lifestyle program.

INTERVENTIONS:
Behavioral: Life style change and weight reduction — Nutritional, behavioural, and exercise counselling to reduce body weight by 10%, normalise blood glucose, lipids, blood pressure, and testosterone level.
  Arms: Intensive treatment group

SUMMARY:
Men diagnosed with metabolic syndrome (MetS) including obesity, hypertension, dyslipidemia and infertility will be assessed for cardiovascular and diabetes risk. The eligible patient will be randomised to one-year life-style intervention program including nutritional, behavioural and exercise counselling or standard care by the general physician. The aim of the program is to reduce cardiovascular and diabetes risks and hypogonadism as well.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years, wish for fatherhood in stable partnership, metabolic syndrome according to guidelines (minimum 3 out of 5 criteria), ready to participate in 1-yr lifestyle program

Exclusion Criteria:

* Not conforming to MetS diagnosis criteria, sterilisation, promiscuous behaviour, contraindications against established medical or surgical treatment of obesity, participation in another weight-loss program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males diagnosed with metabolic syndrome
Enrollment: 70 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with normalisation of diabetes or cardiovascular risk or improvement of hypogonadism | 1 year
  Diabetes risk Glycated hemoglobin >5.7%, Cardiovascular risk score >5%, Hypogonadism score increase of 20 points

CONTACTS AND LOCATIONS:
Locations (1):
- Justus Liebig University, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No